CLINICAL TRIAL: NCT06729476
Title: The Effect of Uroshield on Sputum-specimen Bacterial Growth and Multidrug Resistant Organisms in Mechanically Ventilated Patients
Brief Title: The Effect of Uroshield on Sputum-specimen Bacterial Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0278-15-SZMC
Record Dates: First submitted 2024-12-01; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Mechanically Ventilated Patients
Keywords: tracheostomy; mechanical ventilation; biofilm; sputum culture; multi drug resistant organisms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active device study arm (Active Comparator): Study Procedure: In this study, half of the recruited patients were connected to the UROSHIELD device (study group), while the other half was connected to a similar but inactive sham device (control group). The medical treating team, research team, and the patients themselves were unaware of who received the active device and who was connected to the inactive, sham device. As mentioned, randomization and allocation of devices was performed by a physician not otherwise involved in the conduct of the study or with data processing.
  Interventions: Device: Uroshield vibrator device
- Sham device control arm (Placebo Comparator): Study Procedure: In this study, half of the recruited patients were connected to the UROSHIELD device (study group), while the other half was connected to a similar but inactive sham device (control group). The medical treating team, research team, and the patients themselves were unaware of who received the active device and who was connected to the inactive, sham device. As mentioned, randomization and allocation of devices was performed by a physician not otherwise involved in the conduct of the study or with data processing.
  Interventions: Device: Uroshield vibrator device

INTERVENTIONS:
Device: Uroshield vibrator device — UROSHIELDTM is a small device that generates low-energy surface acoustic waves, which transmit energy to the endotracheal tube through a thin cable attached to the tube. Laboratory studies using catheterized urinary tract models have shown a significant reduction in microbial colonization and reduced development of antimicrobial resistance in UROSHIELDTM device treated individuals.

SUMMARY:
The investigators retrospectively register the conduct of this study after its completion.

DETAILED DESCRIPTION:
Background: Ventilator-associated pneumonia is a frequent complication of mechanical ventilation, caused by bacterial proliferation and biofilm formation on endotracheal tubes. The UROSHIELDTM is a small device that generates low-energy surface acoustic waves, which transmit energy to the endotracheal tube through a thin cable attached to the tube. Laboratory studies using catheterized urinary tract models have shown a significant reduction in microbial colonization and reduced development of antimicrobial resistance in UROSHIELDTM device treated individuals.

Purpose: To evaluate the impact of a UROSHIELDTM device, adapted for endotracheal tube diameter, on the development of positive sputum cultures in intubated patients.

Methods: The study was prospective, double-blind, interventional and randomized. Included were newly intubated patients, who were randomized at a rate of 1:1 by a physician not involved in the study. Patients, treating staff and study investigators were blinded to whether the patients received true or sham devices. Sputum cultures were taken at baseline and every three days for 15 days.

ELIGIBILITY:
Inclusion Criteria:

Mechanically ventilated patients

Exclusion Criteria:

Less than 18 years of age, pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Sputum-specimen bacterial growth | six months
  Sputum specimen collection at day 0 and then every third day for 15 days.
Growth of multidrug resistant organisms from sputum cultures | six months
  Isolation of sputum specimens collected at day 0 and then every third day for 15 days.

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Friedmann, MD, Study Director — Shaare Zedek Medical Center

IPD SHARING:
Plan to Share IPD: No